CLINICAL TRIAL: NCT04788251
Title: Falls Prevention Evaluation and Development for Older Adults in the Community
Acronym: FREDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geriatric Education and Research Institute (Other Government)
Collaborators: Ministry of Health, Singapore (Other Government); Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other); Singapore Institute of Technology (Other); Duke-NUS Graduate Medical School (Other); Monash University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2020/01193
Record Dates: First submitted 2021-01-19; First posted 2021-03-09 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Physical Performance; Fear of Falling
Keywords: Accidental fall; Older adult

STUDY DESIGN:
Intervention Model Description: This is a stepped-wedge cluster randomized trial in which there will be a sequential crossover of clusters from the waitlist control to the intervention period where the sequence of crossover is randomized. The clusters are defined as groups with at least 5 participants. Each of the North and Central regions will have 6 clusters.
  The intervention will be sequentially rolled out to 12 clusters that are randomized to 6 time periods (sequences). Each sequence has 6 steps where one step has a duration of 8 weeks. The intervention will be rolled out sequentially to 2 clusters (1 North, 1 Central) at every step until all 12 clusters have received the intervention by the end of the study. Each cluster will have 1-3 community sites and minimum 5 participants. Outcome assessors will be blinded to sequence allocation.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise-based fall prevention intervention (Experimental): To receive 7 weeks of exercise-based programme
  Interventions: Other: Exercise-based fall prevention intervention (Modified Otago Exercise Programme and Modified Stepping On Programme)
- Wait-list controls (Other): To receive fall prevention resources while waiting for programme
  Interventions: Other: Wait-list control

INTERVENTIONS:
Other: Exercise-based fall prevention intervention (Modified Otago Exercise Programme and Modified Stepping On Programme) — The modified OEP is a group exercise programme that consists of progressive strength and balance exercises led by trained exercise leaders (fitness instructors or health coaches). The supervised sessions will be conducted twice a week (1 hour each) for 7 weeks. Participants will be given an exercise booklet and encouraged to exercise at home.
  The modified SOP is a group fall prevention programme that consists of exercise sessions and discussions on various falls prevention aspects facilitated by a trained programme leader and supported by programme facilitators and peer facilitators. The supervised sessions will be conducted once a week (2 hours each) for 7 weeks. Participants will be given homework and encouraged to exercise at home. In addition, there will be an optional home visit (Week 11), a 1-hour booster session (Week 19) and a telephone call (Week 31).
  Arms: Exercise-based fall prevention intervention
Other: Wait-list control — To receive fall prevention resources while waiting for their programme to start
  Arms: Wait-list controls

SUMMARY:
Exercise-based fall prevention programmes with strength and balance components have been shown to reduce the rate of falls, risk of falling, fractures and injuries. However, there is little evidence on the implementation of these programmes in real-world settings.

This study aims to assess the effectiveness of exercise-based fall prevention interventions on fall risk (physical performance and fear of falling) among community-dwelling older adults who are at risk of falling in Singapore. A secondary aim is to assess the effectiveness of the programme on other health outcomes. The study will also evaluate the programme implementation from 3 perspectives of older adults, implementers and community partners.

DETAILED DESCRIPTION:
Two exercise-based fall prevention programmes (Otago Exercise Programme, OEP and the Stepping On Programme, SOP) have been shown to be effective to prevent and reduce falls in primarily non-Asian settings. The Otago Exercise Programme is a single component intervention that has been shown to reduce fall rate among older adults by 35%. The OEP is a group-based exercise programme based on strength and balance components. The Stepping-On Programme is a multi-component intervention that has been shown to reduce fall rate by 30%. The SOP consists of group-based series of weekly sessions to teach fall prevention strategies to community-dwelling older adults. Sessions comprise of strength-balance exercises and classes based on adult learning principles.

However, there is little evidence of the effectiveness, feasibility and acceptability of locally-adapted community fall prevention interventions. Furthermore, studies on the effectiveness of fall prevention interventions among Asian populations are less robust due to the lack of well-designed studies with adequately powered sample sizes.

In this study, exercise-based fall prevention programmes will be implemented based on geographic region where participants living in the North region will receive the modified SOP and participants in the Central region will receive the modified OEP.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years and above
* Lives in the community
* Living in the Central or North region of Singapore
* Singaporean or Singapore Permanent Resident
* Understand conversational English or Chinese
* Able to walk independently in the community with or without assistive devices (Defined as single-point walking aid, e.g. umbrella, cane, walking stick)
* Answered 'Yes' to any of 3 falls risk screening questions (i.e. 1. Did you have a fall in the past 12 months?, 2. Are you concerned about falling?, 3. Do you feel like you are going to fall when getting up or walking?)

Exclusion Criteria:

* Currently participating in other falls prevention programme or trial or participated in a fall prevention programme or trial in the past 3 months
* Has chest pains when doing exercise
* Had a recent major surgery less than 3 months or is undergoing renal dialysis or active cancer treatment
* Has been told by a doctor to have the following medical conditions: Dementia, Severe neuromuscular or cardiovascular conditions i.e. stroke in the past 6 months, heart failure, acute myocardial infarction, Parkinson's disease
* Have been told by a doctor not to exercise due to health issues
* Score of less than 7 on the Abbreviated Mental Test (AMT)

Ages: 60 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2022-10-29 (Actual)

PRIMARY OUTCOMES:
Difference in Mobility Between Intervention and Control Blocks | Data will be collected at baseline and immediately after each step as this is a stepped-wedge analysis.
  Measured using the Timed Up and Go (TUG)

SECONDARY OUTCOMES:
Difference in Physical Performance Between Intervention and Control Blocks | Data will be collected at baseline and immediately after each step as this is a stepped-wedge analysis.
  Measured using the Short Physical Performance Battery (SPPB). A summary score (range 0-12) will be calculated, with higher score indicating a better performance.
Difference in Fear of Falling Between Intervention and Control Blocks | Data will be collected at baseline and immediately after each step as this is a stepped-wedge analysis.
  Measured using the 16-item Falls Efficacy Scale International (FES-I). The score ranges from 16 to 64, with a higher score indicating a greater fear of falling.

OTHER OUTCOMES:
Falls and Injurious Falls | Data will be collected at baseline and immediately after each step
  Number of falls, rate of falls and number of fall-related injuries will be measured as secondary outcomes. Fall-related health utilization in terms of hospitalization or institutionalization will also be measured.
Subjective Health | Data will be collected at baseline and immediately after each step
  Measured by asking "In general, how would you say your health is?"
Health-Related Quality of Life | Data will be collected at baseline and immediately after each step
  Measured using the 5-level EuroQol 5-dimension (EQ-5D-5L) scales. It will be used to assess health-related quality of life in 5 dimensions, whereby each dimensions will be scored on a 5-point rating scale: no problems, slight problems, moderate problems, severe problems, and extreme problems. Scores will be combined and converted to a single index value.
Fall-Related Protective Behaviours | Data will be collected immediately pre- and post-intervention
  Measured using the revised Falls Behavioural Scale (FaB) that includes 24 statements that describe day-to-day behaviours and actions, both habitual and intentional, that if not done safely, can place an individual at undue risk of falling. Participants will respond with a four-point Likert scale. Higher score indicates safer behaviours.
Loneliness | Data will be collected at baseline and immediately after each step
  Measured using the revised UCLA 3-item Loneliness Scale. The score ranges from 3 to 9, with people from 3-5 as 'not lonely' and people score 6-9 as 'lonely'.
Falls-Related Healthcare Utilization Cost | Data will be collected at baseline and immediately after each step
  Measured using the Client Service Receipt Inventory (CSRI)
Productivity Loss | Data will be collected at baseline and immediately after each step
  Measured using the Work Productivity and Activity Impairment Questionnaire-General Health (WPAI-GH)

CONTACTS AND LOCATIONS:
Overall Officials: Chek Hooi Wong, MBBS, FRCP, MPH, Principal Investigator — Geriatric Education and Research Institute
Locations (2):
- Singapore (2):
  - Tan Tock Seng Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tan PJ, Ginting ML, Lim ZZB, Balachandar N, Sultana R, Kadir MM, Xu T, Ismail NH, Yap JKY, Wong SF, Yoong J, Matchar DB, Hill K, Wong CH. Pragmatic multicentre stepped-wedge cluster randomised trial to investigate the effectiveness of community-based falls prevention programme for older adults with falls risk in Singapore: a protocol paper. BMJ Open. 2023 Jun 1;13(6):e072029. doi: 10.1136/bmjopen-2023-072029. PMID 37263684